CLINICAL TRIAL: NCT05765227
Title: Clinical Evaluation of a Manufacturing Process for a Frequent Replacement Silicone Hydrogel Multifocal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLN705-M103
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Refractive Ametropia
Keywords: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID#224381, then AOHG MF (Other): Lehfilcon A multifocal contact lenses worn first, with lotrafilcon B multifocal contact lenses worn second in pre-determined order. Each study lens type will be worn bilaterally (in both eyes) for approximately 2 days. CLEAR CARE will be used for nightly cleaning and disinfection.
  Interventions: Device: Lehfilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses; Device: Hydrogen peroxide-based cleaning and disinfection system
- AOHG MF, then LID#224381 (Other): Lotrafilcon B multifocal contact lenses worn first, with lehfilcon A multifocal contact lenses worn second in pre-determined order. Each study lens type will be worn bilaterally (in both eyes) for approximately 2 days. CLEAR CARE will be used for nightly cleaning and disinfection.
  Interventions: Device: Lehfilcon A multifocal contact lenses; Device: Lotrafilcon B multifocal contact lenses; Device: Hydrogen peroxide-based cleaning and disinfection system

INTERVENTIONS:
Device: Lehfilcon A multifocal contact lenses — Investigational silicone hydrogel multifocal contact lenses
  Other Names: LID#224381 MF contact lenses
Device: Lotrafilcon B multifocal contact lenses — Commercially available silicone hydrogel multifocal contact lenses
  Other Names: AOHG MF contact lenses; AIR OPTIX® plus HydraGlyde ® multifocal contact lenses (AOHG MF)
Device: Hydrogen peroxide-based cleaning and disinfection system — Commercially available cleaning and disinfection system for silicone hydrogel contact lenses
  Other Names: CLEAR CARE®

SUMMARY:
The purpose of this clinical trial was to evaluate the clinical performance of a manufacturing process on a frequent replacement multifocal contact lens.

DETAILED DESCRIPTION:
Subjects will be expected to attend 3 scheduled visits. Eligible subjects will wear each study lens type in a cross-over fashion for approximately 2 days.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an consent form (ICF) that has been approved by an Institutional Review Board (IRB);
* Willing to stop wearing habitual contact lenses for the duration of study participation;
* Currently wearing multifocal soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Any eye infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator;
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator;
* History of refractive surgery, or plan to have refractive surgery during the study;
* Current or history of dry eye in either eye that would preclude contact lens wear, in the opinion of the investigator;
* Monovision contact lens wear;
* Other protocol-defined exclusion criteria may apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (1):
- Johns Creek Research Clinic, Johns Creek, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 investigative site located in 1 country (US).
Pre-assignment Details: Of the 18 enrolled, 1 participant was exited prior to study start as a screen failure. This reporting group includes all participants exposed to any study lenses evaluated in this study (17).
Groups:
- LID#224381, Then AOHG MF: Lehfilcon A multifocal contact lenses worn first, with lotrafilcon B multifocal contact lenses worn second in pre-determined order. Each study lens type was worn bilaterally (in both eyes) for approximately 2 days in a daily wear modality. CLEAR CARE was used for nightly cleaning and disinfection.
- AOHG MF, Then LID#224381: Lotrafilcon B multifocal contact lenses worn first, with lehfilcon A multifocal contact lenses worn second in pre-determined order. Each study lens type was worn bilaterally (in both eyes) for approximately 2 days in a daily wear modality. CLEAR CARE was used for nightly cleaning and disinfection.
Period: First Wear Period (Approx. 2 Days)
Arm/Group | LID#224381, Then AOHG MF | AOHG MF, Then LID#224381
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0
Period: Second Wear Period (Approx. 2 Days)
Arm/Group | LID#224381, Then AOHG MF | AOHG MF, Then LID#224381
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | LID#224381, Then AOHG MF | AOHG MF, Then LID#224381 | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (4.3) | 62.4 (5.2) | 63.2 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 5 | 8 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 7 | 14
  Black or African American | 1 | 2 | 3
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Binocular Visual Acuity (VA) With Study Lenses at 4 Meters (logMAR)
Description: VA was assessed binocularly (both eyes together) using a letter chart and measured in logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity. No hypothesis testing was prespecified for this endpoint.
Time Frame: Day 2, each study lens type worn during the corresponding crossover period
Population: This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- LID#224381: Lehfilcon A multifocal contact lenses worn during first wear period or second wear period, as pre-determined.
- AOHG MF: Lotrafilcon B multifocal contact lenses worn during first wear period or second wear period, as pre-determined.
Arm/Group | LID#224381 | AOHG MF
Number analyzed (Participants) | 17 | 17
logMAR | -0.08 (0.06) | -0.06 (0.06)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from time of consent to study exit, up to 10 days.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of subjects. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses.
- LID#224381 Ocular; LID#224381 Nonocular: Events reported in this group occurred while exposed to lehfilcon A multifocal contact lenses.
- AOHG MF Ocular; AOHG MF Nonocular: Events reported in this group occurred while exposed to lotrafilcon B multifocal contact lenses.
Arm/Group | Pretreatment | LID#224381 Ocular | LID#224381 Nonocular | AOHG MF Ocular | AOHG MF Nonocular
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/34 | 0/17 | 0/34 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/34 | 0/17 | 0/34 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/34 | 0/17 | 0/34 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT05765227/Prot_SAP_000.pdf